CLINICAL TRIAL: NCT01869686
Title: An Open-label Study to Evaluate the Concentration of Denosumab in Seminal Fluid After a Single Subcutaneous Injection in Healthy Men
Brief Title: Study to Evaluate the Concentration of Denosumab in Seminal Fluid in Healthy Men After a Single Subcutaneous Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 20120351
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental): single subcutaneous injection
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — 60 mg
  Other Names: Prolia (R)

SUMMARY:
This is a phase 1b, open-label, single dose study in healthy male subjects. Approximately 12 healthy male subjects will receive a subcutaneous injection of denosumab on Day 1. Subjects will be followed by a 105 day treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Subject has provided informed consent; Healthy male between ≥40 to ≤ 65 years of age (inclusive) at the time of enrollment; Subject must be willing and able to produce a semen sample on seven separate study visits; Subject must be willing to refrain from ejaculation for a 48 hour period prior to each sample collection;

Exclusion Criteria:

Any condition or drug therapy that might interfere with the subjects ability to ejaculate and produce a semen sample; Clinically significant abnormality during the screening physical examination, ECG, or laboratory evaluation; Known history of blood in urine or semen; Osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (eg, tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal and/or pre-existing dental disease; Recent tooth extraction (within 6 months of screening visit); Evidence of hypocalcemia at screening; Known vitamin D deficiency; Malignancy (except non-melanoma skin cancers) within the last 5 years; Positive for human immunodeficiency virus (HIV) at screening or known diagnosis of AIDS; Positive Hepatitis B Surface Antigen (HepBsAg) (indicative of chronic Hepatitis B) or detectable Hepatitis C virus Ribonucleic acid (RNA) by Polymerase Chain Reaction (PCR) at screening (indicative of active Hepatitis C - screening is generally done by Hepatitis C Antibody (HepCAb), followed by Hepatitis C virus RNA by PCR if HepCAb is positive); History of hypersensitivity or allergic reaction to mammalian cell derived drug products or sensitivity to any of the products or components to be administered during dosing; Known intolerance to calcium or vitamin D supplements; Subject previously has entered this study or has been previously exposed to denosumab in the past 12 months; Has donated or lost ≥ 400 mL of blood or plasma within 8 weeks prior to screening; Positive urine screen for alcohol and/or potential drugs of abuse at screening unless medication is prescribed by a physician and approved by the Investigator and Amgen; Known alcohol abuse or use of illicit drugs within 12 months of enrollment; Subject is unwilling or unable to limit alcohol consumption throughout the course of the study. Alcohol is prohibited 24 hours prior to screening and administration of investigational product. Alcohol is limited to no more than 2 drinks per day for the duration of the study; where a standard drink is equivalent to 12 ounces of regular beer, 8-9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits; Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives (whichever is longer) since ending treatment on another investigational device or drug study(s). Other investigational procedures while participating in this study are excluded; Use of any non-Amgen approved over-the-counter or prescription medications, within the 14 days or 5 half-lives (whichever is longer), prior to receiving the dose of denosumab. Acetaminophen (up to 2 g per day) for analgesia and hormone replacement therapy (eg, androgen, thyroid) will be allowed. Other medications may be approved following review by the Principal Investigator and the Amgen Medical Monitor. Written documentation of this review and Amgen acknowledgement is required for subject participation; Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and Investigator's knowledge; Subject has any kind of disorder that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures; History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 17 June 2013; last patient enrolled 17 June 2013.
Groups:
- Denosumab: Participants received a single subcutaneous injection of 60 mg denosumab on Day 1.
Period: Overall Study
Arm/Group | Denosumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black (or African American) | 0
  Mixed race | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 11
  Othe | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.73 (4.21)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Denosumab in Seminal Fluid
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 12
ng/mL | 100 (81.9)

2. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Denosumab in Seminal Fluid
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population with available data
Measure: Median (Full Range); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 11
days | 21 (81.9) [8.0 to 49]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Denosumab in Seminal Fluid
Description: The area under the denosumab seminal fluid concentration-time curve from time zero to last quantifiable concentration (AUClast), estimated using the linear trapezoidal method.
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 12
days*ng/mL | 5220 (4880) [8.0 to 49]

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Denosumab in Serum
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 12
ng/mL | 6170 (2070)

5. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Denosumab in Serum
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 12
days | 8.0 (81.9) [7.9 to 21]

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Denosumab in Serum
Description: The area under the denosumab serum concentration-time curve from time zero to last quantifiable concentration (AUClast), estimated using the linear trapezoidal method.
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 12
days*ng/mL | 333000 (122000) [8.0 to 49]

7. Secondary Outcome: Ratio of Maximum Seminal Fluid Concentration by the Serum Concentration (Cmax Ratio)
Description: The ratio of maximum denosumab seminal fluid concentration over the denosumab serum concentration at the corresponding time point (Cmax Ratio)
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population with available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Denosumab
Number analyzed (Participants) | 11
ratio | 0.0217 (0.0154) [8.0 to 49]

8. Secondary Outcome: Ratio of Seminal Fluid AUC by Serum AUC for the 106 Day Dosing Period
Description: The ratio of denosumab seminal fluid AUC over denosumab serum AUC for the 106-day dosing period.
Time Frame: Days 1, 10, 22, 36, 50, 78 and 106
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Denosumab
Number analyzed (Participants) | 12
ratio | 0.0170 (0.0148) [8.0 to 49]

9. Secondary Outcome: Ratio of Denosumab Seminal Fluid Concentration Over the Denosumab Serum Concentration at the Last Study Time Point (Day 106).
Time Frame: Day 106
Population: Pharmacokinetic population with available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Denosumab
Number analyzed (Participants) | 11
ratio | 0.0197 (0.0318) [8.0 to 49]

ADVERSE EVENTS:
Time Frame: 78 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Denosumab 60 mg SC
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60 mg SC (N=12)
Vertigo positional (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60 mg SC (N=12)
Rectal haemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.